CLINICAL TRIAL: NCT06560541
Title: A Randomized and Open Label Phase 2 Clinical Trial of Low-GI, Polyphenol-Rich UKMRC9 Red Rice on Cardiometabolic Parameters in Patients With Type 2 Diabetes
Brief Title: Rice Intervention in Chronic Health Study
Acronym: RICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taylor's University (Other)
Collaborators: National University of Malaysia (Other); Universiti Putra Malaysia (Other); National Institutes of Health, Ministry of Health Malaysia (Other); University of Nottingham Malaysia (Other)
Responsible Party: Principal Investigator, Tilakavati Karupaiah, Professor, Taylor's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD0120Q1410
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pigmented rice; Whole grain rice; Type 2 diabetes; Cardio-metabolic health; Mitochondrial DNA methylation; Circulating exosomal miRNA; Metabolomics; Consumer acceptance test
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: Although the participants will not be blinded to the investigator product (IP), they will be masked from the brand of the IP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diabetes Patients Cohort Red Rice (DPC-RR) (Experimental)
  Interventions: Other: UKMRC9
- Diabetes Patients Cohort White Rice (DPC-WR) (Placebo Comparator)
  Interventions: Other: White rice
- Healthy Control Cohort Red Rice (HCC-RR) (Experimental)
  Interventions: Other: UKMRC9
- Healthy Control Cohort White Rice (HCC-WR) (Placebo Comparator)
  Interventions: Other: White rice

INTERVENTIONS:
Other: UKMRC9 — UKMRC9 is a low glycemic index and polyphenol-rich red pigmented rice
  Arms: Diabetes Patients Cohort Red Rice (DPC-RR); Healthy Control Cohort Red Rice (HCC-RR)
Other: White rice — White rice refers to a local polished rice
  Arms: Diabetes Patients Cohort White Rice (DPC-WR); Healthy Control Cohort White Rice (HCC-WR)

SUMMARY:
The goal of this clinical trial is to learn if the low glycemic index (GI), polyphenol-rich red pigmented rice (UKMRC9) works to improve cardio-metabolic parameters in Malaysian adults with type 2 diabetes (T2D) and healthy individuals. It will also learn about the molecular and metabolic effects of UKMRC9 as well as its consumer acceptance. The main questions it aims to answer are:

1. What are the effects of substituting white rice with UKMRC9 on cardio-metabolic parameters, including adiposity indices, glycemic control, lipid profiles, appetite hormones, total antioxidant capacity, inflammatory markers, blood pressure, and 10-year cardiovascular risk in Malaysian adults T2D patients and healthy individuals?
2. What are the effects of substituting white rice with UKMRC9 on urinary and plasma metabolome in Malaysian adults T2D patients and healthy individuals?
3. What are the effects of substituting white rice with UKMRC9 on mitochondrial DNA methylation and circulating exosomal microRNAs expression in Malaysian adults T2D patients and healthy individuals?
4. What is the difference in consumer acceptance toward UKMRC9 compared to white rice?
5. What are the facilitators and barriers to the inclusion of UKMRC9 as a staple food in Malaysian diet?
6. What are the dietary quality and dietary pattern among Malaysian adults T2D patients and healthy individuals?
7. What is the effects of substituting white rice with UKMRC9 on advanced glycation end (AGE) products among Malaysian adults T2D patients and healthy individuals?

Researchers will compare UKMRC9 to white rice to see if UKMRC9 works to improve cardio-metabolic parameters in Malaysian adults T2D patients and healthy individuals.

Participants will:

* Take UKMRC9 or white rice everyday for 24 weeks.
* Visit the study sites once every 12 weeks for follow-up assessments.
* Share their experience in substituting white rice with UKMRC9 in focus group discussion at the end of the intervention.

ELIGIBILITY:
Diabetes Arm:

Inclusion Criteria:

* Attending outpatient clinics
* Age 18 - 60 years (i.e. adult population)
* Both male and female
* Regular consumption of polished white rice (presumably high-GI) ≥ 200g/day
* Established T2DM patients on oral medication
* Glycated hemoglobin (HbA1c) 7% to 10%
* Willing to take part and being compliant to the study protocol

Exclusion Criteria:

* Glycated hemoglobin (HbA1c) <7% or >10%
* Use of insulin
* A change in the type of treatment (e.g. insulin injection) during the intervention period
* Regular consumption of low-GI rice types (basmati) or colored rice (red rice, purple rice, black rice) for ≥3 months.
* Oral corticosteroids > 3 months
* Pregnancy
* Unstable medical condition.
* Undergone any major operation in the past 3 months
* Chronic alcohol drinker.
* Not on weight loss diets or supplementation.
* Taking part in another clinical trial.

Healthy arm:

Inclusion Criteria:

* Healthy free living
* With glycated haemoglobin (HbA1c <6.3%)
* Age 18 - 60 years (i.e. adult population)
* Both male and female
* Regular consumption of polished white rice (presumably high-GI) ≥ 200g/day
* Generally, physically and mentally healthy as per medical examination.
* Willing to take part and being compliant to the study protocol.

Exclusion Criteria:

* Regular consumption of low-GI rice types (basmati) or colored rice (red rice, purple rice, black rice) for ≥3 months
* Presence of gastrointestinal disease, metabolic diseases such as diabetes, kidney failure, liver or pancreatic disease, hyperthyroidism, cancer or severe malnutrition.
* Oral corticosteroids > 3 months
* Pregnancy
* Undergone any major operation in the past 3 months
* Chronic alcohol drinker.
* Not on weight loss diets or supplementation..
* Taking part in another clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Changes in cardio-metabolic parameters | Baseline versus 12-week versus 24-week
  Effects of UKMRC9 on cardio-metabolic parameters including adiposity indices, glycemic control, lipid profiles, appetite hormones, total antioxidant capacity, inflammatory markers, blood pressure, and 10-year cardiovascular risk
Changes in urinary and plasma metabolome | Baseline versus 12-week versus 24-week
  Effects of UKMRC9 on urinary and plasma metabolome
Changes in mitochondrial DNA methylation and circulating miRNAs expression | Baseline versus 24-week
  Effects of UKMRC9 on mitochondrial DNA methylation and circulating miRNAs expression

SECONDARY OUTCOMES:
Consumer Acceptance Test | Baseline versus 12-week versus 24-week
  Difference in consumer acceptance between UKMRC9 and white rice
Facilitators and Barriers to the Inclusion of UKMRC9 as a staple food | 24-week
  Participants' experience of substituting white rice with UKMRC9 explored through the focus group discussions.
Dietary Pattern of Malaysian Adults with and without diabetes | Baseline screening
  The dietary pattern will be assessed at baseline using two distinct methods to provide a comprehensive evaluation of dietary intakes: (1) 3-day diet record, which will capture short-term food intakes and (2) food frequency questionnaire, which assess habitual, long term dietary intakes. The dietary data from each method will be reported in gram per day (g/d) and analysed separately using dimension reduction techniques to produce unified dietary pattern scores. This score will be categorized into tertiles (T1: 0-33.3%, T2: 33.4-66.7%, T3: 66.8-100%) for further analysis. Higher tertile indicates stronger adherence to the established dietary pattern.
Diet Quality of Malaysian Adults with and without diabetes | Baseline screening
  Diet quality will be benchmarked using the Healthy Eating Index (ranging from 0 to 100%), where a higher index indicates better diet quality.
Changes in Advanced Glycation End (AGEs) products measured by skin autofluorescence using AGE Reader mu (Diagnostics). | Baseline versus 12-week versus 24-week
  This outcome measure assesses the effects of UKMRC9 on the levels of advanced glycation end products (AGEs) as measured by skin autofluorescence, using the AGE Reader mu (Diagnostic). The results will be expressed in arbitrary units (AU)

CONTACTS AND LOCATIONS:
Overall Officials: Tilakavati Karupaiah, PhD, Principal Investigator — Taylor's University
Locations (10):
- Malaysia (10):
  - Hospital Canselor Tuanku Muhriz, Cheras, Kuala Lumpur
  - Klinik Kesihatan Cheras, Cheras, Kuala Lumpur
  - Klinik Kesihatan Bandar Baru Bangi, Bangi, Selangor
  - Klinik Kesihatan Kajang, Kajang, Selangor
  - Klinik Kesihatan Sungai Chua, Kajang, Selangor
  - The University of Nottingham Malaysia Compus, Semenyih, Selangor
  - Hospital Pengajar Universiti Putra Malaysia, Seri Kembangan, Selangor
  - Universiti Putra Malaysia, Seri Kembangan, Selangor
  - Institute for Medical Research, Shah Alam, Selangor
  - Taylor's University, Subang Jaya, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu J, Balaji B, Tinajero M, Jarvis S, Khan T, Vasudevan S, Ranawana V, Poobalan A, Bhupathiraju S, Sun Q, Willett W, Hu FB, Jenkins DJA, Mohan V, Malik VS. White rice, brown rice and the risk of type 2 diabetes: a systematic review and meta-analysis. BMJ Open. 2022 Sep 27;12(9):e065426. doi: 10.1136/bmjopen-2022-065426. PMID 36167362
- [Background] Golzarand M, Toolabi K, Eskandari Delfan S, Mirmiran P. The effect of brown rice compared to white rice on adiposity indices, lipid profile, and glycemic markers: a systematic review and meta-analysis of randomized controlled trials. Crit Rev Food Sci Nutr. 2022;62(27):7395-7412. doi: 10.1080/10408398.2021.1914541. Epub 2021 Apr 27. PMID 33905269
- [Background] Abdul Rahim AF, Norhayati MN, Zainudin AM. The effect of a brown-rice diets on glycemic control and metabolic parameters in prediabetes and type 2 diabetes mellitus: a meta-analysis of randomized controlled trials and controlled clinical trials. PeerJ. 2021 May 26;9:e11291. doi: 10.7717/peerj.11291. eCollection 2021. PMID 34123581
- [Background] Mendoza-Sarmiento D, Mistades EV, Hill AM. Effect of Pigmented Rice Consumption on Cardiometabolic Risk Factors: A Systematic Review of Randomized Controlled Trials. Curr Nutr Rep. 2023 Dec;12(4):797-812. doi: 10.1007/s13668-023-00496-7. Epub 2023 Sep 7. PMID 37676476
- [Background] Malik VS, Sudha V, Wedick NM, RamyaBai M, Vijayalakshmi P, Lakshmipriya N, Gayathri R, Kokila A, Jones C, Hong B, Li R, Krishnaswamy K, Anjana RM, Spiegelman D, Willett WC, Hu FB, Mohan V. Substituting brown rice for white rice on diabetes risk factors in India: a randomised controlled trial. Br J Nutr. 2019 Jun;121(12):1389-1397. doi: 10.1017/S000711451900076X. Epub 2019 Apr 22. PMID 31006420